

Provider Skill Building for Engagement and Communication in Healthcare – Hypertension Management (REACH – Hypertension)

#### **CONCISE SUMMARY**

**Purpose of the Study:** This research aims to evaluate the effectiveness of an intervention designed to enhance primary care clinicians' skill in talking to, listening to, and working with their patients.

**Initial Assessments:** At the beginning of the study, clinician participants will be asked to complete three surveys.

**Patient Involvement:** Clinician participants will be asked to provide consent for their patients to participate in the study and to audio record their clinical visit. **Clinician Intervention:** The intervention consists of six 30-minute sessions,

including three learning modules and three coaching sessions.

**Study Duration:** The study will last approximately 6-8 months. This includes 6-12 weeks to complete the intervention and periodic audio recordings of your clinical encounters.

There is a risk of loss of confidentiality. There is a possible benefit of improving your skills in patient-centered care.

If you are interested in learning more about this study, please continue to read below.

Research studies are voluntary. You do not have to agree to be in this study. Please read this consent form carefully and take your time making your decision. The study team will discuss the study with you. Please ask about any words or information that you do not clearly understand. We encourage you to talk with your family and friends before you decide to take part in this research study. The nature of the study, risks, inconveniences, discomforts, and other important information about the study are listed below and will be reviewed with you by the study team.

Please tell the study doctor or study staff if you are taking part in another research study.

Dr. Sarah Wilson and Dr. Laura Svetkey will conduct the study. The study is funded by a grant from National Institutes of Health (NIH) / National Heart, Lung,



Provider Skill Building for Engagement and Communication in Healthcare – Hypertension Management (REACH – Hypertension)

and Blood Institute (NHLBI). Portions of Sarah Wilson and Laura Svetkey and their research team's salaries will be paid by this grant.

### Why is this study being done?

The purpose of this study is to increase clinicians' skills in talking to, listening to, and working with their patients. We will look at how clinicians interact with diverse populations.

### How many people will take part in this study?

Approximately 20 clinicians and 150 patients from Duke University Medical Center will take part in this study.

### What is involved in the study?

If you agree to participate in this study, you will need to sign and date this consent form. You will also be asked to complete a baseline survey, which includes your date of birth, gender identity, race and ethnicity, clinical specialty, years in practice, and practice characteristics (such as work schedule, number of patients, and self-reported communication style).

All participants will receive the intervention – because this is an early stage of research, there is no control group. Before starting the intervention, you will complete two Implicit Association Tests (IATs). One test focuses on race, and the other on race adherence. You will take these tests using a secure, confidential link through Project Implicit, a safe and secure platform for collecting data on implicit social cognition. The results will only be accessible to you and the study personnel for research or analysis purposes.

The intervention consists of six, 30-min curriculum activities including three learning modules that can be completed on your own and three one-on-one virtual coaching sessions. The study will last approximately 6-12 weeks, depending on whether you complete the six sessions weekly or bi-weekly.

Both, before the intervention and at two follow-up timepoints after the intervention, we will enroll 2-3 of your patients and ask them to audio-record their clinical visit with you. We will ask you to allow us to send a letter from you to patients scheduled to see you during each patient recruitment period. Patients who do not "opt out" will be contacted by study staff before a scheduled visit with you.



## ADULT: Clinician Consent Form Provider Skill Building for Engagement and Communication

Provider Skill Building for Engagement and Communication in Healthcare – Hypertension Management (REACH – Hypertension)

If they choose to participate, study staff will meet them in the waiting room on the day of the visit to complete enrollment and instruct them on audio recording procedures. Audio recording will involve the patient bringing a pre-programmed tablet into the exam room to record all that is said by you or them during the visit. The recordings will be confidential and used by study personnel only.

After the clinical visit, we will ask your patients to complete a follow-up survey.

### How long will I be in this study?

After you complete the baseline survey and IATs using Project Implicit (a safe and secure platform for collecting data on implicit social cognition), we will collect baseline audio recorded clinical visits with your enrolled patients. These baseline assessments and 2-3 audio recorded clinical visits will occur within 1-2 weeks after signing the consent. After the baseline assessments and audio recordings, you will begin the intervention which will last about 6-12 week. After you complete the intervention, we will recruit 2-3 patients scheduled for visits with you at 2-6 weeks and 2-3 patients scheduled for visits with you at 12-16 weeks to audio record those encounters. Therefore, you will be enrolled in the study for approximately 6-8 months.

Participation is voluntary. You can choose to stop participating at any time without penalty or loss of any benefits to which you are entitled.

### What are the risks of the study?

There are no physical risks with being in this study. There is, however, the potential risk of loss of confidentiality. Every effort will be made to keep your information confidential. However, this cannot be guaranteed. We will email you a copy of this consent form; however, email is not a secure method of communication. By signing this consent form and providing your email, you agree that we may email you a copy of this consent form. We will be using Project Implicit to administer the two Implicit Association Tests (IATs) - Race and Race-Adherence. Project Implicit is a safe and secure platform for collecting data on implicit social cognition. To complete the IATs, you will sign into a secure confidential link to Project Implicit. Data exchanged with this site are protected by SSL encryption. Project Implicit uses the same secure hypertext transfer protocol (HTTPS) that banks use to transfer credit card information securely. This provides strong security for data transfer to and from the website. IP addresses are



Provider Skill Building for Engagement and Communication in Healthcare – Hypertension Management (REACH – Hypertension)

routinely recorded but are completely confidential. Results will only be available to you and study personnel. If your encounters are audio recorded with your permission, the recordings will be stored electronically on a password protected, encrypted computer that will be kept in a locked office at Duke University. The recordings will not be shared with anyone outside of the research team. Once the study is complete, the audio recordings will be destroyed. Some of the questions we will ask you as part of this study may make you feel uncomfortable. You may refuse to answer any of these questions, and you may take a break at any time during the study. You may stop your participation in this study at any time.

### **Unforeseeable Risks:**

While we do not have any unforeseeable risks to disclose, there may be risks that are not yet known.

### Are there benefits to taking part in the study?

If you agree to take part in this study, there are no direct medical benefits to you. We hope the information learned from this study will benefit providers in this study and patients and providers in the future.

### Will my information be kept confidential?

Participation in research involves some loss of privacy. We will do our best to make sure that information about you is kept confidential, but we cannot guarantee total confidentiality. Your personal information may be viewed by individuals involved in this research and may be seen by people including those funding, and regulating the study, and those currently collaborating on the study and those who will possibly be collaborating on the study in the future. We will share only the minimum necessary information in order to conduct the research. Your personal information may also be given out if required by law. The Department of Health and Human Services (HHS) has issued a Certificate of Confidentiality to further protect your privacy. With this Certificate, the investigators may not disclose research information that may identify you in any Federal, State, or local civil, criminal, administrative, legislative, or other proceedings, unless you have consented for this use. Research information protected by this Certificate cannot be disclosed to anyone else who is not connected with the research unless:



# Consent to Participate in a Research Study ADULT: Clinician Consent Form Provider Skill Building for Engagement and Communication in Healthcare - Hypertension Management (REACH - Hypertension)

- 1) there is a law that requires disclosure (such as to report child abuse or communicable diseases but not for legal proceedings);
- 2) you have consented to the disclosure, including for your medical treatment; or
- 3) the research information is used for other scientific research, as allowed by federal regulations protecting research subjects.

Disclosure is required, however, for audit or program evaluation requested by the agency that is funding this project.

You should understand that a Confidentiality Certificate does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it. This means that you and your family must also actively protect your own privacy.

We will be using Project Implicit (a safe and secure platform for collecting data on implicit social cognition) to administer the two Implicit Association Tests (IATs) - Race and Race-Adherence. To complete the IATs, you will sign into a secure confidential link to Project Implicit. Data exchanged with this site are protected by SSL encryption. Project Implicit uses the same secure hypertext transfer protocol (HTTPS) that banks use to transfer credit card information securely. This provides strong security for data transfer to and from the website. IP addresses are routinely recorded but are completely confidential. Results will only be available to you and study personnel.

Finally, you should understand that the investigator is not prevented from taking steps, including reporting to authorities, to prevent serious harm to yourself or others.

The study results will be retained in your research record for at least six years after the study is completed. At that time either the research information not already in your medical record may be destroyed or information identifying you will be removed from such study results at DUHS. Any research information in your medical record will be kept indefinitely.



Provider Skill Building for Engagement and Communication in Healthcare – Hypertension Management (REACH – Hypertension)

This information may be further disclosed by the sponsor of this study. If disclosed by the sponsor, the information is no longer covered by federal privacy regulations. If this information is disclosed to outside reviewers for audit purposes, it may be further disclosed by them and may not be covered by federal privacy regulations.

While the information and data resulting from this study may be presented at scientific meetings or published in a scientific journal, your name or other personal information will not be revealed.

Some people or groups who receive your health information might not have to follow the same privacy rules. Once your information is shared outside of DUHS, we cannot guarantee that it will remain private. If you decide to share private information with anyone not involved in the study, the federal law designed to protect your health information privacy may no longer apply to the information you have shared. Other laws may or may not protect sharing of private health information

### **Certificate of Confidentiality:**

The National Institutes of Health (NIH) / National Heart, Lung, and Blood Institute (NHLBI) has issued a Certificate of Confidentiality (CoC) for this study. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or lawsuit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings, like a court order.

There are some important things that you need to know about the CoC:

It DOES NOT stop reporting required by federal, state or local laws. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others.

It CANNOT BE USED to stop a sponsoring United States federal or state

DUHS RB
IRB NUMBER: Pro00115680
IRB REFERENCE DATE: 04/23/2025
IRB EXPIRATION DATE: 08/01/2026



Provider Skill Building for Engagement and Communication in Healthcare – Hypertension Management (REACH – Hypertension)

government agency from checking records or evaluating programs, including when the Food and Drug Administration (FDA) requires it.

It DOES NOT prevent your information from being used for other research if allowed by federal law.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other people not connected with the study. The CoC does not stop you from willingly releasing information about your involvement in this study. It also does not prevent you from having access to your own information.

### Will it cost me anything to be in the study?

There are no additional costs to you for participating in this study. You and your insurance company will not be billed for your participation.

### Will I be paid to be in the study?

You will be provided with a meal in the clinic or receive a restaurant voucher for all curriculum sessions (total of 6 meals or vouchers). You will receive continuing education (CE) credit for completing the intervention (i.e. learning modules and coaching sessions).

### What if I want to withdraw from the study?

If you agree to be in the study, you may withdraw from the study at any time. If you withdraw from the study, no new data about you will be collected for study purposes other than data needed to keep track of your withdrawal.

Your decision not to participate or to withdraw from the study will not involve any penalty or loss of benefits to which you are entitled, and will not affect your access to health care at Duke. Also, nonparticipation or withdrawal from this study will not affect your job status if you are a Duke employee and will not affect your grades if you are a Duke student.

Additionally, we will tell you about new information that may affect your health, welfare, or willingness to stay in this study.



Provider Skill Building for Engagement and Communication in Healthcare – Hypertension Management (REACH – Hypertension)

The use of your data and samples may result in commercial profit. You will not be compensated for the use of your data and samples other than what is described in this consent form.

### Registration on the web site ClinicalTrials.gov:

A description of this clinical trial will be available on <a href="https://clinicaltrials.gov/">https://clinicaltrials.gov/</a> as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### Whom should I call if I have questions or problems?

For questions about the study or a research-related injury, or if you have problems, concerns, questions or suggestions about the research, contact Dr. Wilson at 919-971-2406 or Dr. Svetkey at 919-819-0238 either during regular business hours or after hours and on weekends and holidays.

You can call the Duke University Health System Institutional Review Board (IRB) Office at (919) 668-5111 if:

- You have question about your rights as a research participant
- You wish to discuss problems related to the research
- You have any concerns or suggestions related to the research
- Want to obtain information or offer input about the research

Form M0345



Consent to Participate in a Research Study ADULT: Clinician Consent Form

 $P_{\underline{r}}$ ovider Skill Building for  $\underline{E}$ ngagement  $\underline{a}$ nd  $\underline{C}$ ommunication in  $\underline{H}$ ealthcare – Hypertension Management (REACH – Hypertension)

### STATEMENT OF CONSENT

"The purpose of this study, procedures to be followed, risks and benefits have been explained to me. I have been allowed to ask questions, and my questions have been answered to my satisfaction. I have been told whom to contact if I have questions, to discuss problems, concerns, or suggestions related to the research, or to obtain information or offer input about the research. I have read this consent form and agree to be in this study, with the understanding that I may withdraw at any time. I have been told that I will be given a signed and dated copy of this consent form."

| Signature of Participant Signature of Person Obtaining Consent | Date | Time |
|---|---|---|
| | <br>Date | <br>Time |